CLINICAL TRIAL: NCT06306027
Title: The Effect of Web-Based Education Program Applied to The Patients Undergoing Knee Arthroplasty on Self-Care Power, Self-Efficacy, and Quality of Life
Brief Title: The Impact of Web-Based Education on Self-Care Power, Self-Efficacy, and Quality of Life in Knee Arthroplasty Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Serap Sayar, Assistant Professor, PhD, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2023/024
Record Dates: First submitted 2024-02-02; First posted 2024-03-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthroplasty
Keywords: Web-Based Education; Self-Efficacy; Quality of Life; Self Care Power; Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): When patients come to the polyclinic for a check-up 15 days after discharge, the web-designed training program site will be promoted. The patient who accepts the research will be given a user name and password specifically created by the researcher. The patient will be explained practically how to log in to the system at home via phone. Patients will be asked to watch educational videos on the website at least twice a week for one month. Then, pre-test data, Personal Information Form, Self-Efficacy Scale, Self-Care Power Scale and Quality of Life Scale data will be collected. Patients who receive training for a month will be asked to fill out the self-efficacy scale, self-care power scale and quality of life scale for post-test data via the mobile application at the end of the month.
  Interventions: Behavioral: Web-based education
- Control Group (No Intervention): When patients come to the outpatient clinic for a check-up 15 days after discharge, they will be asked to fill out the Personal Information Form, Self-Efficacy Scale, Self-Care Ability Scale, and Quality of Life Scale by face-to-face information collection method.Patients will receive routine treatment, care and checks in line with the institutional policy. A web designed training program will not be implemented. One month after the pre-test data is collected, patients will be called and asked to fill out the self-efficacy scale, self-care ability scale and quality of life scale when they come to the outpatient clinic.

INTERVENTIONS:
Behavioral: Web-based education — The patient discharged after knee arthroplasty surgery will attend a follow-up appointment 15 days later, and during this visit, they will be granted permission to resume work. The patient will receive detailed information about accessing, entering, and using the web-based training. Scales with pre-test data will be completed by the patient. They will be encouraged to log in at least twice a week, and the patient will be monitored for a total of 1 month (4 weeks). After one month, the patient will be asked to fill out the scales again.
  Arms: Experimental

SUMMARY:
The knee joint, which we use actively every day, is the largest joint in our body that bears the weight, allowing various movements such as walking, running, squatting, and standing. It involves the largest load-bearing structures in the body, including bones, cartilage, surrounding muscles, and ligaments, facilitating the mobilization of the joint. Due to constant use, the knee joint is susceptible to injuries and wear. Total knee arthroplasty (TKA) surgery involves replacing a degenerated joint surface, often due to conditions like osteoarthritis or rheumatoid arthritis, with a metal or polyethylene prosthesis. TKA, a widely used and highly successful surgical intervention in recent years, reduces pain, enhances functional range of motion, and improves independence and quality of life. Severe pain following TKA surgery restricts the movement of the knee joint and daily life activities, leading to the patient's inadequacy in self-care. Patients undergoing TKA surgery often face a lack of information after discharge. This lack of knowledge, coupled with uncertainty about the disease, limits the patient's self-efficacy. As the self-care power diminishes for patients struggling with daily life activities, their self-efficacy is negatively affected. The continuity of education becomes crucial since the verbal and written instructions given after surgery may not be sustained, causing a gradual decline in an individual's self-efficacy. As seen in the literature, studies have shown that postoperative pain, swelling, joint stiffness, fear, and movement limitations negatively impact the quality of life for patients undergoing TKA. Consequently, the self-care capacity, self-efficacy levels, and quality of life for individuals who have undergone TKA are adversely affected, as indicated in the literature.Ensuring continuity of care at home is crucial not only during the early postoperative period in the clinic but also after discharge. The nurse plays a significant role as an educator/advisor after discharge. The nurse provides counseling to patients discharged after Total Knee Arthroplasty (TKA) on pain management, disease progression, rehabilitation process, exercises, and considerations during daily activities (such as walking, bathing, toileting). Additionally, the nurse offers guidance on late-stage complications that may arise at home due to surgery and situations requiring hospitalization. While web-based educational interventions have been conducted for various patient groups, a web-based education program specifically for TKA surgery has not been identified. Having web-based post-TKA patient education allows continuous monitoring, assesses attendance and effectiveness remotely, and enables individuals to convey requests and questions to researchers through live support, ultimately enhancing the effectiveness of education. This approach is believed to prevent complications, reduce patient care costs and readmissions, increase patients' self-sufficiency in self-care, and consequently elevate their self-efficacy levels and quality of life. Close monitoring of postoperative patients is expected to improve their quality of life and self-care abilities, leading to increased satisfaction with healthcare services.

DETAILED DESCRIPTION:
The knee joint, actively used every day, is the largest joint in our body, supporting the body's weight and enabling various movements such as walking, running, squatting, and standing. It involves the most load-bearing structures: bones (distal femur, proximal tibia, and patella), cartilage (meniscus and articular cartilage), surrounding muscles, and ligaments (infrapatellar fat pad), facilitating joint mobilization. Due to constant use, the knee joint is prone to injuries and wear, making it the most common site for Osteoarthritis (OA). In the treatment of knee OA, conservative measures, medical treatments, and physical therapy are utilized in the early stages. However, when these treatments are ineffective, arthroplasty surgery, a commonly used surgical method, is often employed. Total Knee Arthroplasty (TKA) involves replacing a degenerated joint surface (femoral, tibial, and patellar joints) with a metal or polyethylene prosthesis. TKA, a widely used and highly successful surgical intervention in recent years, reduces pain, enhances functional range of motion, and improves independence and quality of life. Although TKA is a successful surgical treatment method, it can also lead to postoperative complications and undesired situations in patients. Post-TKA, patients often require support and information to regain their previous independence, especially since severe postoperative pain restricts knee joint movement and daily life activities, leading to insufficient self-careLiterature indicates that patients undergoing Total Knee Arthroplasty (TKA) experience adverse effects on their self-care power, self-efficacy levels, and quality of life. In this context, nurses, who are primarily responsible for patient care, have significant duties. Besides early postoperative care in the clinic, ensuring the continuity of home care after discharge is crucial. It has been reported in the literature that the care needs of discharged patients continue at home, and patients require high levels of education to safely continue their lives with a joint prosthesis. After discharge, the nurse's role as an educator/advisor becomes crucial. The nurse provides detailed counseling to patients discharged after TKA. The education provided by nurses enables patients to adapt to living with a joint prosthesis and actively participate in decisions related to their own care. With advancements in information technology, patient education has transitioned to the web using devices such as phones, tablets, and computers. Web-based education is advantageous due to constant access to information and the provision of continuous education through written and visual materials.As seen in the literature, web-designed educational studies have been conducted on different patient groups, but no web-designed educational study has been found after TKA surgery. Having a web design for post-TKA patient education will increase the effectiveness of the training, as patients can be tracked at any time, the effectiveness of the training can be measured remotely, whether they attend the training or not, and the researcher can send their requests and questions via live support, thus preventing possible complications, reducing patient care costs and re-use. It is thought that it will reduce hospitalizations, increase the self-care power of patients by becoming self-sufficient, and therefore increase their self-efficacy levels and quality of life. It is predicted that patients' satisfaction with health care services will increase as their quality of life and self-care abilities will increase when they are closely monitored one-on-one after the surgery.

ELIGIBILITY:
Inclusion Criteria:

Being 18 years or older

* First time performing Total Knee Arthroplasty
* Ability to access the internet via smart phone, tablet, computer
* Must have the ability to use smart phones and tablets
* Ability to read and understand Turkish
* No mental, psychiatric or neurological disability

Exclusion Criteria:

* Complications develop in the patient during the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 1 Minutes
  The personal information form has been created by researchers based on a literature review. This form includes a total of 14 questions covering sociodemographic and introductory characteristics of the patient, such as age, gender, weight, height, BMI, marital status, education level, occupation, employment status, cohabitants, presence of chronic diseases, regularly used medications, and the status of receiving discharge education.

SECONDARY OUTCOMES:
Self-Care Power Scale | 3 Minutes
  The Self-Care Power Scale is designed to measure an individual's ability to take care of themselves or assess their capabilities. The scale consists of 35 items, each rated on a five-point Likert scale ranging from 0 to 4. Scores on the scale range from a minimum of 0 to a maximum of 140, with higher scores indicating an increase in self-care power. The Cronbach's Alpha value for the scale is 0.92.

OTHER OUTCOMES:
Self-Efficacy - Competence Scale | 2 Minutes
  The Self-Efficacy-Competence Scale is a Likert-type self-assessment scale designed to evaluate behavior and behavioral changes. The highest possible score on the scale is 115, and the lowest is 23. A higher total score on the scale indicates a high general perception of self-efficacy and competence, while a lower total score suggests a low perception of self-efficacy and competence. The Cronbach's alpha coefficient for the scale is 0.81.
Short Form 36 Quality of Life Scale | 4 Minutes
  Short Form 36 Quality of Life Scale is designed to assess the quality of life. The reliability coefficient (α-Cronbach) of the scale ranges between 0.73 and 0.76. The scale consists of 8 subscales related to health, totaling 36 items. Separate total scores are provided for each subscale, with scores ranging from 0 to 100. A decrease in scores from the scale indicates poor quality of life, while an increase suggests good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Serap SAYAR, PhD, Study Director — KTO Karatay University; Esra Nur BOZTAŞ, MScN, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researcher at Konya City Hospital will collect the data.